CLINICAL TRIAL: NCT02258737
Title: Efficacy of Transitional Case Management Following Psychiatric Hospital Discharge: a Randomized Trial
Brief Title: Efficacy of Transitional Case Management Following Psychiatric Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Charles Bonsack, Professor, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMT
Record Dates: First submitted 2014-09-29; First posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Mental Disorders
Keywords: Case management; psychiatric hospitalization; discharge
MeSH Terms: conditions — Mental Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- transitional case management (Experimental)
  Interventions: Behavioral: Transitional Case Management
- standard care (Active Comparator)
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Transitional Case Management — The case management activity deals with organizational and clinical aspects. The objective is to focus on network's expectations during hospitalization and at discharge, and ensure contacts between hospital and patient' social network. The aim is to support patient during the transition phase following discharge
  Arms: transitional case management
Behavioral: Standard Care — Routine hospitalization care is broadly defined as the usual level of care in the context of the adult department of psychiatry of the CHUV (Centre Hospitalier Universitaire Vaudois).
  Arms: standard care

SUMMARY:
Efficacy of transitional case management following psychiatric hospital discharge: a randomized trial

Background The movement of deinstitutionalisation in Western societies has modified the role of psychiatric hospital, which has lost its asylum function to become a place for acute care.

Psychiatric stays are now shorter and close interactions with the outpatient care network is therefore more critical than before. The first weeks following discharge from psychiatric hospital represent a period of high risk for relapse, readmission or even suicide. Case management has a proven efficacy in facilitating patients' deinstitutionalisation after very long hospitalisations and in stabilizing high users of psychiatric care. In contrast, studies exploring the impact of time limited case management following discharge from short stays (transitional case management) in earlier phases of psychiatric disorders in connection with primary care are lacking.

Working Hypotheses The investigators hypothesize that transitional case management following hospital discharge decreases risk of readmission, improves adherence to outpatient care, facilitates recovery and improves patients' satisfaction with treatment as compared to routine care.

Specific Aims In this study, the investigators will compare the impact of both intervention on number of contact and level of adherence to outpatient care. The investigators will also compare both groups on number of readmission, risk of early aggravation of the disorders, level of functioning and satisfaction with care.

Methods This is a randomized single-blind study comparing transitional case management after discharge with routine post-hospitalization care for subjects living independently without institutional psychiatric follow-up. Demographic and clinical data will be gathered during hospitalization, and 1, 3, 6 and 12 months after discharge. Quantitative assessment of outcomes using validated instruments will be: contact and level of adherence to outpatient care (primary outcomes), as well as number of hospitalization days, number of readmissions, severity of illness and satisfaction with care (secondary outcomes).

Expected Value of the Proposed Project This study should improve psychiatric patients follow-up in collaboration with the different levels of care in the global context of deinstitutionalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18-65 years of age
* No immediate institutional follow up after discharge
* Independent living condition

Exclusion Criteria:

* Organic brain disease
* Clinically significant concurrent illnesses
* Poor understanding of French

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Adherence to outpatient care | one year
  Information on admission, diagnoses, notes on problems of compliance, preparation for hospital discharge and links with outpatient care using the Boyer Scale (Boyer, McAlpine, Pottick et al. 2000)
Working alliance | one year
  Assessment of the relationship between patient and care provider uning the Working Alliance Inventory, short version (WAI-SRp) (Horvath, 1984; Hatcherr & Gillaspy, 2006; translation : Baillargeon & Leduc, 2000; de Roten, 2006)
Number of readmissions | one year
  Socio-demographic assessment of service receipt (use of services, length of hospitalization and number of readmissions) and medication profile using the Client Socio-Demographic and Service Receipt Inventory (CSSRI - EU) (Chisholm et al., 2000)
Degree of psychiatric symptoms | one year
  Assessment of psychiatric symptoms (global severity, diversity of symptoms and degree of discomfort) using the Symptom check-list (SCL-90 R) (Derogatis, 1977; French translation: Guelfi et Dreyfus,1984)
Hopelessness | one year
  Assessment of the risks of suicide attempts or of suicide. Assessment of pessimism using the Hopelessness Scale - Questionnaire H (Hopelessness scale) (Beck, 1974; translation Cottraux, 1985)
Substance use | one year
  Assessment of alcohol and drug consumption (prevalence and frequency) using an extract from " Cannabis and Substance Use Assessment Scale " (CASUAS) (Edwards et al., 2003)
Perceived Improvement | one year
  Assessment of the patient's perception of clinical improvement using the Perceived Improvement questionnaire (Perreault, 2003)
Severity of mental health problems | one year
  Assessment of the severity of mental health problems (behavior, handicap, symptoms, social) using the Health of Nation Outcome Scale (HoNOS) (Wing & Curtis, 1996; Lauzon et al. 2001)
Global Assessment of Functioning | one year
  Assessment of the patient's level of global functioning on a scale of 0 to 100 using the Global Assessment of Functioning (GAF), (Endicott, Spitzer et al 1976; translation Guelfi, Boyer, 1989)
Social and Occupational Functioning | one year
  Assessment of the levels of social and professional functioning on a scale of 0 to 100 using the Social and Occupational Functioning Assessment Scale (SOFAS) (Goldman, Skodol et Lave, 1992)
Social support | one year
  Assessment of the network's and of the patient's perception regarding availability using the " Social Support " questionnaire (Community Mental Health Evaluation Initiative, CMHEI, 2001)
Empowerment | one year
  Measure of empowerment using the "Empowerment" questionnaire (Community Mental Health Evaluation Initiative, CMHEI, 2001)
Satisfaction | one year
  Assessment of the degree of satisfaction of users of psychiatric services using the Client's Satisfaction Questionnaire (CSQ- 8) (Larsen, 1979; translation Chambon, 1992)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bonsack, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Social Psychiatry Section, Lausanne University Hospital, Prilly, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Bonsack C, Golay P, Gibellini Manetti S, Gebel S, Ferrari P, Besse C, Favrod J, Morandi S. Linking Primary and Secondary Care after Psychiatric Hospitalization: Comparison between Transitional Case Management Setting and Routine Care for Common Mental Disorders. Front Psychiatry. 2016 Jun 2;7:96. doi: 10.3389/fpsyt.2016.00096. eCollection 2016. PMID 27313547